CLINICAL TRIAL: NCT03643809
Title: Epidemiology and Clinico-genetic Correlations of Auto-inflammatory Diseases
Brief Title: Epidemiology of SAIDs.
Acronym: EPIMAI
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0368
Record Dates: First submitted 2018-07-26; First posted 2018-08-23 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Autoinflammatory Diseases
Keywords: Systemic autoinflammatory diseases (SAIDs)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Systemic autoinflammatory diseases (SAIDs) are inflammatory conditions caused by a defect of the innate immune system. Most are hereditary, but little is known on recent entities. The investigators aim to (1) establish correlations between the main mutations and symptoms presented by patients (genotype-phenotype correlation), and (2) describe the most recently described clinical, genetic, and demographic characteristics of SAIDs.

DETAILED DESCRIPTION:
Background SAIDs are a heterogeneous group of diseases linked to a deregulation of the innate immune system. They are characterized by systemic or organ inflammatory attacks. In the absence of accurate diagnosis and adequate treatment, evolution can be lethal. Most SAIDs are hereditary, and the diagnosis is based on genetic analysis because the clinical features overlap. The investigators have been among the first in France to routinely develop Next Generation Sequencing (NGS), which allows a simultaneous and exhaustive analysis of a constantly evolving panel of now more than 60 genes involved in SAIDs. While there are epidemiological studies on the first described MAIs, nothing has been done regarding the newest clinical entities.

Objectives The investigators want to study and value the data the investigators have collected on the most recent SAIDs (500 patients) Main objective: Establish correlations between the main mutations and symptoms presented by patients (genotype-phenotype correlation).

Secondary objectives: Descriptive epidemiology study: Describe the most recently described clinical, genetic, and demographic characteristics of SAIDs.

Methodology The investigators have over the last 20 years set up a database that continues to evolve. These data are collected prospectively from patients (N> 7000) with SAID refered to our laboratory for genetic analysis. This database contains invaluable demographic, clinical and genetic data, carefully collected for each patient, on a standard file of analysis request made with clinicians from the reference center for auto-inflammatory diseases and amyloidosis (CeRéMAIA). The collection of consent is systematic (declared collection).

ELIGIBILITY:
Inclusion Criteria:

- NGS autoinflammatory panel performed

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred to the laboratory for suspected systemic autoinflammatory diseases (SAID)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-07-07 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Number of genetically ascertained patients | 1 day
  Number of genetically ascertained patients

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume SARRABAY, Principal Investigator — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, Montepllier, France